CLINICAL TRIAL: NCT00061477
Title: ALIMTA Plus Gemcitabine as Front-Line Chemotherapy for Patients With Malignant Pleural or Peritoneal Mesothelioma: A Phase II Clinical Trial
Brief Title: Pemetrexed Plus Gemcitabine as Front-Line Chemotherapy for Patients With Malignant Pleural or Peritoneal Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7214; H3E-US-JMFZ; NCT00060190 (obsolete NCT alias)
Record Dates: First submitted 2003-05-28; First posted 2003-05-29 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Pemetrexed; Gemcitabine

INTERVENTIONS:
Drug: Pemetrexed
Drug: Gemcitabine

SUMMARY:
The purposes of this study are to determine:

1. The safety of Pemetrexed plus Gemcitabine and any side effects that might be associated with the combination of these two drugs.
2. Whether Pemetrexed plus Gemcitabine can help patients with mesothelioma live longer.
3. Whether Pemetrexed plus Gemcitabine can make the tumor smaller or disappear, and for how long.
4. To see if patients feel better while taking Pemetrexed plus Gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mesothelioma that can be treated with chemotherapy
* Have received no prior chemotherapy for mesothelioma
* Have at least one measurable lesion
* Have an adequate performance status
* Sign an informed consent

Exclusion Criteria:

* Previous treatment with chemotherapy for mesothelioma
* Treatment with an investigational drug within the last 30 days, previously completed or withdrawn from this study or any other study investigating Pemetrexed
* Treatment with radiation therapy within the last 4 weeks
* Brain metastasis that is uncontrolled
* Active infection or other serious condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2002-12; Study Completion 2006-09

PRIMARY OUTCOMES:
To determine the objective tumor response rate for pemetrexed plus gemcitabine every 21 days in patients with malignant pleural mesothelioma who have not received prior chemotherapy

SECONDARY OUTCOMES:
To assess time to objective tumor response for responding patients;To assess duration of response for responding patients;To assess time to treatment failure;To assess time to progressive disease
To assess progression-free survival;To assess overall survival;To determine toxicities of pemetrexed in combination with gemcitabine in this population

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania